CLINICAL TRIAL: NCT02826967
Title: Feasibility and Effectiveness of Colonic Irrigation as a Non-oral, Same-day Bowel Preparation Option in Patients Undergoing Screening or Surveillance Colonoscopy
Brief Title: Feasibility and Effectiveness of Colonic Irrigation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 institutional restrictions on screening colonoscopies
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-00578
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Colonic Irrigation
Keywords: Hydro-San Plus colonic irrigation system; Screening colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Colonic Irrigation (Experimental): A designated health professional will administer to the patient the colonic irrigation procedure -using the Hydro-San Plus colon therapy system, an FDA approved and ISO certified device for colonic irrigation and cleansing before endoscopic procedures (FDA #2027347).
  Interventions: Procedure: Colonic Irrigation

INTERVENTIONS:
Procedure: Colonic Irrigation

SUMMARY:
This study will allow investigators to determine whether colonic irrigation may allow for a non-oral, same-day alternative to traditional oral bowel prep regimens. This in turn could lead to more persons able to undergo screening colonoscopy for colorectal cancer and thus increased cancer prevention and early detection.

DETAILED DESCRIPTION:
The primary endpoints for this study are:

* Overall quality of bowel cleansing for each of the three segments of the colon (ascending, transverse, and descending) as measured by the Boston Bowel Preparation Score (BBPS), a validated numerical scale for bowel cleanse (0-3 for each colon segment; 0-9 total score) (6).
* Patient satisfaction, as measured by a questionnaire administered by a study investigator via follow-up phone call after completion of the colonic irrigation and subsequent colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients age 50-84 years old, who require a screening or surveillance colonoscopy
* Ability to give consent

Exclusion Criteria:

* Pregnancy
* History of ulcerative colitis or Crohn's disease
* History of surgical ostomy
* History of colorectal surgery

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-06; Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Overall quality of bowel cleansing for each of the three segments of the colon (ascending, transverse, and descending) as measured by the Boston Bowel Preparation Score (BBPS) | 15 Minutes
  Boston Bowel Preparation Score (BBPS), a validated numerical scale for bowel cleanse (0-3 for each colon segment; 0-9 total score)
Patient satisfaction, as measured by a questionnaire administered by a study investigator via follow-up phone call after completion of the colonic irrigation and subsequent colonoscopy. | 15 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pochapin, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States